CLINICAL TRIAL: NCT03764553
Title: Liposomal iRInotecan, Carboplatin or oXaliplatin in the First Line Treatment of Esophagogastric Cancer: a Randomized Phase 2 Study
Brief Title: Liposomal iRInotecan, Carboplatin or oXaliplatin for Esophagogastric Cancer
Acronym: LyRICX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_256
Record Dates: First submitted 2018-10-29; First posted 2018-12-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer
Keywords: palliative chemotherapy; metastatic esophagogastric cancer; Efficacy; toxicity
MeSH Terms: conditions — Esophageal Neoplasms | interventions — irinotecan sucrosofate; Carboplatin; Capecitabine; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposomal irinotecan, leucovorin and 5FU (Experimental): IV Nal-IRI 80 mg/m² (expressed as irinotecan hydrochloride (HCl) salt), folinic acid 400 mg/m², fluorouracil 2400 mg/m² over 46 h, every 2 weeks.
  No addition of nivolumab is possible for this arm
  Interventions: Drug: Liposomal Irinotecan; Drug: 5-fluorouracil; Drug: Leucovorin
- Carboplatin and capecitabine (Experimental): IV and PO Capecitabine 1000 mg/m2 and carboplatin area under the curve (AUC5), every three weeks.
  In case of PD-L1 CPS ≥5 only: nivolumab, dose according to local standard, iv day 1
  Interventions: Drug: Carboplatin; Drug: Capecitabine
- oxaliplatin and capecitabine (Experimental): IV and PO Capecitabine 1000 mg/m2 and oxaliplatin 130 mg/m2, every three weeks.
  In case of PD-L1 CPS ≥5 only: nivolumab, dose according to local standard, iv day 1
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Liposomal Irinotecan — Iv liposomal irinotecan
  Arms: Liposomal irinotecan, leucovorin and 5FU
Drug: Carboplatin — IV Carboplatin
  Arms: Carboplatin and capecitabine
Drug: Capecitabine — PO Capecitabine
  Other Names: Xeloda
  Arms: Carboplatin and capecitabine; oxaliplatin and capecitabine
Drug: Oxaliplatin — IV Oxaliplatin
  Arms: oxaliplatin and capecitabine
Drug: 5-fluorouracil — IV 5-fluorouracil
  Arms: Liposomal irinotecan, leucovorin and 5FU
Drug: Leucovorin — IV Leucovorin
  Arms: Liposomal irinotecan, leucovorin and 5FU

SUMMARY:
This is a multi-center, open label, randomized phase II trial for patients with previously untreated metastatic or locally advanced esophagogastric cancer, using a pick the winner design to identify the best combination therapy in terms of progression free survival and neurotoxicity.

DETAILED DESCRIPTION:
The sample size to identify the best combination therapy is based on the following decision making strategy. With less or even zero neurotoxicity grade 2-4 (defined as worst toxicity), the Nal-IRI plus 5FU/LV combination is expected to outperform the standard combination capecitabine plus oxaliplatin and may also outperform capecitabine plus carboplatin. To compensate for a higher neurotoxicity grade 2-4 level, the capecitabine combinations should demonstrate increased progression free survival (PFS) according to the next schedule.

With the addition of nivolumab in the second quarter of 2022, the capecitabine combinations are expected to have a PFS benefit over the Nal-IRI of 0.65 months (50% of the 1.7 months seen in the CM6495, because 50% of the capecitabine regimens will be treated with nivolumab)

If the difference in the percentage of patients experiencing neurotoxicity grade 2-4 stays within the 10-30% range, an increase of at least 3.65 months of PFS identifies the most preferable combination strategy; if the percentage is ≤10% and the PFS increase <3.65 months, but in favor of carboplatin, then the choice should be based on other grade 3-4 toxicities observed; otherwise, the strategy with the lowest level of neurotoxicity grade 2-4 is the most preferable one. At least 4.65 months PFS should be gained to compensate for a difference in neurotoxicity grade 2-4 within the >30 to 50% range.

The total number to be included will be 272. Patients will first be tested for PD-L1 and then will be conditionally randomized. Patients with a PD-L1 CPS <5 or a contraindication for nivolumab treatment, will be randomized to respectively the Nal-IRI plus 5FU, the capecitabine plus carboplatin and capecitabine plus oxaliplatin group following a 2:1:1 scheme. Patients with a PD-L1 CPS ≥5 will be randomized to the capecitabine plus carboplatin and capecitabine plus oxaliplatin group following a 2:1 scheme and will receive nivolumab in addition to chemotherapy treatment.

Taking into account 15% withdrawal of patients from the trial before start of study medication, we will include 320 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent according to International Conference on Harmonization (ICH)/Guideline for Good Clinical practice (GCP), and national/local regulations prior to any screening procedures.
* Male or female adult patients (> 18 years).
* Patients with histologically confirmed diagnosis of metastatic or irresectable human epidermal growth (HER2) negative adenocarcinoma of the stomach or oesophagus; patients with HER2 positive disease are eligible when treatment with trastuzumab is contraindicated. If histology cannot be obtained, cytology is acceptable to prove metastatic disease.
* Patients with metastatic or irresectable adenocarcinoma of the stomach or oesophagus not pre-treated with chemotherapy or radiotherapy for irresectable or metastatic disease. Palliative radiotherapy on the primary tumor or a metastatic lesion is allowed if other untreated lesions eligible for evaluation are present.
* Measurable disease as assessed by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) (WHO) performance status 0-2
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute Neutrophil Count (ANC) > 1.5 x 109 /L
  * Hemoglobin (Hgb) > 5.6 mmol/L
  * Platelets > 100 x 109 /L
* Serum total bilirubin within ≤ 1.5 x ULN (upper limit of normal); or total bilirubin < 3.0 x upper limit of normal (ULN) with direct bilirubin within normal range in patients with well documented Gilbert's syndrome; biliary drainage is allowed for biliary obstruction
* Serum creatinine < 1.5 x ULN or creatinine clearance >30 mL/min/1.73 m2
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 2.5x ULN within normal range or < 5.0 x ULN if liver metastases are present
* If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test, beta-human chorionic gonadotropin (β-hCG) documented 72 hours prior to the first administration of study drug. If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator during the period of administration of study drug and after the end of treatment as recommended.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria:

* Prior systemic treatment for metastatic or irresectable stomach or oesophageal cancer.
* Evidence of disease progression within six months after completion of adjuvant or neoadjuvant treatment (whichever is last) containing a fluoropyrimidine and/or platinum compound and/or irinotecan; progression on neoadjuvant chemoradiation with carboplatin area under the curve (AUC2) and paclitaxel 50 mg/m2 within this time frame is allowed.
* All target lesions in a radiation field without documented disease progression. 11
* Patient has known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
* Past or current malignancy other than entry diagnosis interfering with prognosis of metastatic esophagogastric cancer.
* Known uncontrollable hypersensitivity or contraindications to any of the components of liposomal irinotecan (Nal-IRI) other liposomal irinotecan formulations, irinotecan, fluoropyrimidines, leucovorin, oxaliplatin, carboplatin. Patients with previous dose reductions or delays are eligible.
* Complete dihydropyrimidine dehydrogenase deficiency .
* Patient has active, uncontrolled bacterial, viral or fungal infection(s) requiring systemic therapy.
* Patient has known past or active infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Signs of interstitial lung disease (ILD)
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate patient participation in the clinical study.
* Use of other investigational drugs within 30 days of enrollment.
* Patient is enrolled in any other clinical protocol or investigational trial that will interfere with the primary endpoint.
* Patients who in the investigators' opinion may be unwilling, unable or unlikely to comply with requirements of the study protocol.
* Current use or any use in last two weeks of strong cytochrome P4503A (CYP3A-enzyme), CYP2C8, and/or strong UDP glucuronosyltransferase (UGT1A) inhibitors/inhibitors
* Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use a reliable method of birth control, during therapy and for 3 months following the last dose of study treatment.
* Treatment within 4 weeks with dihydropyrimidine dehydrogenase (DPD) inhibitors, including sorivudine or its chemically related analogues such as brivudine.
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 42 months
  To compare the progression free survival
Number of participants with treatment-related Neurotoxicity | 42 months
  Number of participants with treatment-related Neurotoxicity according to CTCAE v4.0

SECONDARY OUTCOMES:
Overall survival | 54 months
  To determine the overall survival of F-Nal-IRI, capecitabine/Carboplatin (CapCar) and capecitabine/oxaliplatin (CapOx)
response rate | 42 months
  To determine the response rate of F-Nal-IRI, CapCar and CapOx
adverse events | 42 months
  To determine the adverse events of F-Nal-IRI, CapCar and CapOx according to NCI common toxicity criteria (CTC) version 4
Quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ C30)) | 42 months
  Overall Quality of life ranging from 0-100 with 100 being best Quality of Life
percentage subsequent treatment lines | 42 months
  The percentage of patients proceeding to subsequent lines of treatment after progression and describe the types of treatment.
the reasons for forgoing subsequent treatment | 42 months
  Reasons for forgoing subsequent treatment after progression on first-line treatment

OTHER OUTCOMES:
Tumor micro environment | 54 months
  Percentage of stroma and tumor immune infiltrate in metastatic tumor tissue as predictor of response to treatment and survival.
Stromal markers in blood | 54 months
  Concentration of ADAM12 in blood
Growth velocity of patient derived tumor organoids | 54 months
  Growth velocity of tumor organoids after treatment measured in days
ctDNA | 54 months
  Concentration circulating tumour DNA (ctDNA) as a marker of response to treatment
Fecal microbiome | 54 months
  Composition of the fecal microbiome as a potential biomarker for response to treatment and toxicity
Costs associated with treatment of F-Nal-IRI, CapCar and CapOx | 54 months
  The cost effectiveness in terms of QUALYs associated with treatment of F-Nal-IRI, CapCar and CapOx
Stromal Markers in tumor | 54 months
  Expression of ADAM12 in metastatic tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, MD, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (34):
- Netherlands (34):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Ziekenhuisgroep Twente, Almelo
  - Flevoziekenhuis, Almere Stad
  - Meander MC, Amersfoort
  - Academic Medical Center, Medical Oncology, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Nij Smellinghe, Drachten
  - Ziekenhuis Gelderse Vallei, Ede
  - Catherina Ziekenhuis, Eindhoven
  - Treant Zorggroep, Emmen
  - Zuyderland Medisch Centrum, Geleen
  - Admiraal de Ruijter Ziekenhuis, Goes
  - Sint Jansdal, Harderwijk
  - Elkerliek ziekenhuis, Helmond
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Treant zorggroep, Hoogeveen
  - Dijklander ziekenhuis, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilherlmina ziekenhuis, Nijmegen
  - Radboud Universitair Medisch Centrum, Nijmegen
  - VieCurie, Roermond
  - Laurentius Ziekenhuis, Roermond
  - Bravis ziekenhuis locatie Roosendaal, Roosendaal
  - Ikazia ziekenhuis, Rotterdam
  - Maasstadziekenhuis, Rotterdam
  - Rivierenland Ziekenhuis, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - UMCU, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03764553/SAP_001.pdf